CLINICAL TRIAL: NCT07098598
Title: Diagnostic Efficacy of 18F-FAPI-74 PET/CT in Patients With Pancreatic Cancer
Brief Title: Pancreatic Cancer Diagnosis With FAPI-PET Imaging
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Panca-FAPI
Record Dates: First submitted 2025-05-27; First posted 2025-08-01 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-05

CONDITIONS: Positron Emission Tomography; Pancreatic Cancer; FAPI; Diagnostics; Recurrent Pancreatic Cancer; Oncologic Surgery; Imaging, Diagnostic; Staging
MeSH Terms: conditions — Pancreatic Neoplasms; Disease | interventions — Positron Emission Tomography Computed Tomography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Staging (Experimental)
  Interventions: Device: PET/CT

INTERVENTIONS:
Device: PET/CT — PET/CT with FAPI-74 tracer is performed.

SUMMARY:
Staging pancreatic cancer (PC) presents a clinical challenge. Triphasic whole body CT is the primary imaging method in diagnosing, staging and during follow up. Conventional PET/CT with 18F-labelled fluorodeoxyglucose (18F-FDG) has its limitations and therefore has a secondary role in imaging pancreatic cancer patients. These conventional imaging methods are good in detecting primary tumors and distant metastasis but poor in detecting local lymph node metastasis. A new PET tracer, fibroblast activation protein inhibitor (FAPI), targets FAP, a protein overexpressed in cancer-associated fibroblasts. It presents a potential new PET imagining tool.

The objective of this prospective diagnostic study is to evaluate the diagnostic efficacy of 18F-FAPI-74 PET/CT in patients with PC. The aim is to evaluate the sensitivity and specificity of 18F-FAPI-74 in detection of local lymph node metastasis and distant metastasis in patient level in patients with PC in primary staging and when suspected recurrence. 100 patients with PC are enrolled on whom PET/CT studies are performed with the novel 18F-FAPI-74 tracer. The data will be collected between 2024-2026.

ELIGIBILITY:
Inclusion Criteria:

* Suspected primary or recurrent pancreatic cancer
* Subjects must be male or female aged 18-85 years.
* WHO performance score 0-2.
* Subjects must be able and willing to give written informed consent and to comply with the requirements of this study protocol.

Exclusion Criteria:

* Vulnerable study subjects such as described in Finnish law clinical studies (disabled, children, pregnant or breast-feeding women, prisoners) will not be included.
* Study subject is not able to understand the purpose of the study.
* Medical conditions prohibiting whole-body PET/CT imaging.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-10-09 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
1) To assess the sensitivity and specificity of 18F-FAPI-74 PET/CT in detection of local lymph node metastasis in patient level in patients with primary pancreatic cancer | 2 years
2) To assess the sensitivity and specificity 18F-FAPI-74 PET/CT in detection of distant metastasis in patient level in patients with primary pancreatic cancer | 2 years
3) To assess the sensitivity and specificity of 18F-FAPI-74 PET/CT in detection of local lymph node metastasis and distant metastasis in patient level in patients with recurrent pancreatic cancer | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Saila Kauhanen, docent, Principal Investigator — University of Turku and Turku University Hospital
Locations (1):
- Turku PET Centre, Turku University Hospital, Turku, Finland

IPD SHARING:
Plan to Share IPD: No